CLINICAL TRIAL: NCT05804396
Title: The SP-303 PERL Study - Combined Occipital and Trigeminal Nerve Stimulation (eCOT-NS) for Preventive Treatment of Migraine
Brief Title: Combined Occipital and Trigeminal Nerve Stimulation (eCOT-NS) for Preventive Treatment of Migraine
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Neurolief Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP-303-PERL
Record Dates: First submitted 2023-03-26; First posted 2023-04-07 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Active stimulation (Experimental): Relivion® device- Active stimulation
  Interventions: Device: Relivion®

INTERVENTIONS:
Device: Relivion® — Active stimulation device

SUMMARY:
The PERL Study will evaluate the safety and efficacy of a self-administered preventive treatment for migraine headache using combined occipital and trigeminal nerve stimulation (Relivion®).

This is a prospective, non-randomized, single arm, multi-center study designed to evaluate the use of Relivion® in reducing the frequency of headache days against a sham performance goal.

DETAILED DESCRIPTION:
The study will include the following study visits & phases:

* Visit 1 Screening
* Run-in (Baseline) Period - Daily migraine headache diary.
* Visit 2 Enrollment -Study enrollment, device and regimen training.
* Treatment Period- Relivion® migraine preventive treatment for 12 consecutive weeks. Patients will be required to fill in a daily migraine diary.
* Visit 3 Follow Up Visit.
* Visit 4 Follow Up Visit.
* Visit 5 End of study.

After completion of visit 5 the subject's participation will be over.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18 years of age and older.
2. Subject meets the ICHD-3 (2018) diagnostic criteria for either Episodic migraine (<15 headache (HA) days/month) or Chronic (at least 15 days of HA/month with at least 8 days/month migraine days (migraine with and without aura) for > 3 months).
3. Subject migraine age of onset <50 years of age.
4. History of 6 to 24 headache days on average per month for the 3 months preceding study enrolment (based on participant report).
5. Completed at least 21 out of 28 days in the eDiary during run-in period. Partially completed data for the run-in period will be adjusted to reflect an estimated number of days with the outcome of interest per 28-day interval by using the formula (28/x)*y, where x is the number of days with observed data per 28-day period and y is the number of observed days with the outcome of interest.
6. Subject reports 6-24 headache days per 28 days, confirmed by 28 days or adjusted 28 days baseline diary.
7. Subjects on prophylactic migraine treatment are permitted to remain on 1 medication with possible migraine-prophylactic effects if the dose has been stable for at least 3 months prior to the screening visit, and the dose is not expected to change during the course of the study.
8. Subject is willing to and capable of complying with the specified study requirements, provided written Informed Consent can complete the electronic diaries, and can be contacted by telephone.

Exclusion Criteria:

1. Initiating or changing the type, dosage, or frequency of any medications for other indications than migraine that are determined to potentially interfere with the study.
2. Failure on ≥2 well-conducted preventive treatments. A treatment failure (lack of efficacy) trial is characterized as a Level A or Level B evidence-based preventive treatment (medications or a MAB or preventive gepant) for migraine preventive trial taken for a minimum of 2 months, at a minimally adequate dose, that produced less than 50% improvement in MMD reduction). Failure to tolerate a preventive treatment does not constitute a preventive treatment failure.
3. History of other chronic headache conditions such as Chronic tension-type headache, Medication Overuse Headache, New Daily Persistent Headache, and Cluster Headache in the prior 6 months.
4. Use of opiates or barbiturates medications in the prior 3 months.
5. Received parenteral infusions for migraine within the previous 2 weeks.
6. Subject has known uncontrolled epilepsy.
7. History of neuro-interventional procedures such as nerve blocks (within the last month), Botulinum Toxin (within the last 3-months), neurosurgical interventions in the head or neck, or implanted/wearable neurostimulators, electronic devices in the head, cardiac pacemaker, surgical clips above the shoulder line or medical pumps, except for dental implants.
8. Current drug abuse or alcoholism.
9. Subjects participating in other clinical trials evaluating experimental treatments or procedures.
10. Skin lesion, scars, or inflammation in the region of the stimulating electrodes.
11. Personality or somatoform disorder.
12. Pregnancy or Lactation.
13. Women of reproductive age not using a reliable contraceptive method, as determined by the Investigator (NOTE: Females of childbearing potential must have a negative pregnancy test).
14. Documented history of cerebrovascular event.
15. Subject with a recent history of traumatic brain injury (TBI), defined as a disruption in the normal function of the brain that can be caused by a bump, blow, or jolt to the head, or penetrating head injury, within 3 months of study enrollment.
16. Subjects who demonstrate or have a history of any cognitive disorder or impairment, memory loss, dementia, confusion or delirium that, in the opinion of the Investigator, may compromise the integrity of the study data or impact the ability of the subject to comply with the study requirements.
17. Subject diagnosed with other chronic pain disorder which in the opinion of the Investigator may compromise the integrity of the study data or impact the ability of the subject to comply with the study requirements.
18. The subject does not have the basic cognitive and motor skills needed to operate a smartphone.
19. Subject with head circumference smaller than 51 centimeters or head circumference larger than 60 centimeters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11-24 (Actual); Primary Completion 2024-11-24 (Actual); Study Completion 2024-11-24 (Actual)

PRIMARY OUTCOMES:
Mean change in Monthly Migraine Days (MMD). | 3 months
  Mean change from baseline (M0) in Monthly Migraine Days (MMD) comparing with the last 28 treatment days (M3: weeks 9-12).

SECONDARY OUTCOMES:
Proportion of responder subjects | 3 months
  Proportion of responder subjects defined as the percent of subjects achieving at least 50% reduction from baseline (M0) in their monthly migraine days comparing with the last 28 treatment days (M3: weeks 9-12).
Mean change in monthly acute anti-migraine headache drug days. | 3 months
  Mean change in baseline (M0) monthly acute anti-migraine headache drug days comparing with the last 28 treatment days (M3: weeks 9-12).
Mean change total headache days. | 3 months
  Mean change in baseline (M0) total headache days comparing with the last 28 treatment days (M3: weeks 9-12)

CONTACTS AND LOCATIONS:
Overall Officials: Stewart J Tepper, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center

IPD SHARING:
Plan to Share IPD: No